CLINICAL TRIAL: NCT01730326
Title: The Comparison of the Effectiveness of Intravenous Dexketoprofen and Paracetamol in the Treatment of Headache Caused by Acute Migraine Attack in Emergency Service
Brief Title: Intravenous Dexketoprofen and Paracetamol in the Treatment of Headache Caused by Acute Migraine Attack
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Mustafa Serinken, Pamukkale University denizli / TURKEY, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: turkcuer 001
Record Dates: First submitted 2012-11-05; First posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Acute Migraine
Keywords: Headache; paracetamol; dexketoprofen; emergency department
MeSH Terms: conditions — Headache; Emergencies | interventions — Acetaminophen; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol (Experimental): Paracetamol which will be given after randomization will be diluted in serum physiologic and will be given as intravenous rapid infusion.
  Interventions: Drug: Paracetamol
- Dexketoprofen (Active Comparator): Dexketoprofen which will be given after randomization will be diluted in serum physiologic and will be given as intravenous rapid infusion.
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Paracetamol — 1000 mg
  Other Names: perfalgan 10 mg/ml
  Arms: Paracetamol
Drug: Dexketoprofen — 50 mg
  Other Names: arveles 50 mg/2 ml
  Arms: Dexketoprofen

SUMMARY:
Patients with acute migraine attack make up the majority of patients consulting the emergency services due to headache. The aim of treatment in the emergency service is to achieve a minimum level of undesirable side effects and to quickly relieve the pain which will not repeat after discharge from the emergency service. Ideal drug treatment contraindication should be at a minimum level and not trigger migraine. Paracetamol and Nonsteroidal anti-inflammatory drugs are often used in the treatment of migraine headache.

Although narcotic analgesics provide effective and rapid analgesia, they have such side effects as hypotension, nausea and vomiting, drowsiness. In recent years, with the production of parenteral forms of non-steroidal anti-inflammatory painkillers, the analgesic efficacy of these drugs has been one of the topics of interest to researchers. Especially intravenous form of paracetamol is new yet compared to other Nonsteroidal anti-inflammatory drugs, and it is a drug with a wide safety margin and less incidence of side effects. The effectiveness of the Intravenous form of paracetamol and whether it can be an alternative to other analgesics is one of the major research topics today, and more study is needed on this subject.

Both drugs are often used in emergency services to treat headache caused by acute migraine attack. Our aim is to compare the effectiveness of intravenous dexketoprofen with paracetamol in the treatment of the headache caused by acute migraine attack.

DETAILED DESCRIPTION:
Materials and Methods of Research:

Among the patients consulting the emergency service with a complaint of headache, those who meet the criteria of 'International Classification of Headache Disorders criteria for migraine without aura' and agreed to participate in the study will form the study group.

The patients forming the study group will be included in the study after they are evaluated according to the criteria of inclusion or exclusion. Our research is an equivalence study. Provided that the difference between the groups is 50 %, α: 99 %, and 1-β: 80 %, it has been determined that each group should include at least 94 subjects, and the number of voluntary subjects has been determined as 200, each group containing 100 subjects.

First of all, in the measurement of the frequency of headaches, the standard 11-point Numeric Rating Scale (NRS), whose reliability is proven, and 100-mm visual analog scale (VAS) will be used. For NRS, patients will be asked to score their pain on a scale ranging from 0 to 10, scoring 0 (zero) in the absence of pain, and 10 in the case of most severe pain; whereas, for VAS, they will be asked to score their pain on a scale ranging from 0 to 100, scoring 0 in the absence of pain, and 100 in the case of most severe pain. Verbal rating scale (VRS) with 4 standard points will be used as another measurement tool. In this measurement, patients will be asked to express their pain as severe, moderate, mild and no pain.

The patients will be divided to two groups.

Groups and drug doses to be given;

1. group: Dexketoprofen Trometamol (50 mg)
2. group: Paracetamol (1000 mg)

The drug which will be given after randomization will be diluted in 150 ml serum physiologic and will be given as intravenous rapid infusion.

The pains of the patients will be assessed in 0., 15. and 30. minutes by NRS, VAS and VRS, and they will be monitored for vital signs and possible side effects.

In 30. minute, the study will be ended, and If the pain continues, fentanyl 1 mcg / kg will be given.

When a patient eligible for the study consults, after obtaining the patient's written consent, the patient will be assigned to one of the study groups based on the next study number. Randomization of study numbers will be prepared by someone other than a person working in the emergency service with the help of a computer, and until the completion of the study, which number is assigned to which drug will be known only by that person. One of the nurses working in the emergency department will be responsible for preparing the study drug, while the other nurse blindly will be responsible for giving the study drug. The numbers belong to the previously enumerated study groups will be stored in envelopes which do not show the inside (allocation concealment), and the study drug will be prepared after the next envelope is opened by the study nurse. Patients eligible for the study will be taken to the unit called 'observation with monitor' in the emergency department, monitored and IV vascular access will be established. The study drugs will be prepared by the emergency nurse responsible for the study and will be given by the other nurse. Medicines prepared for each group are transparent and same.

ELIGIBILITY:
1. Inclusion Criteria:

   a. Patients who are 18 years of age and older, and who agreed to participate in the study will be included in the study.
2. Exclusion Criteria:

   1. Patients having received analgesic in the last six hours,
   2. pregnant women,
   3. women of childbearing potential and not using birth control,
   4. those who do not agree to participate in the study,
   5. those under age of 18, those who have signs of peritoneal irritation,
   6. those who are allergic to drugs used in the study,
   7. hemodynamically unstable patients,
   8. patients with renal transplant,
   9. those who suffer from liver, kidney, cardiac and pulmonary insufficiency and others with systemic diseases,
   10. patients with vision problems and those who are illiterate will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Reduction in visual analogue scale and Numeric Rating Scale | 15 minutes interval
  The pain of the study subjects was measured after 15th and 30th minutes later after the study drug administered.

SECONDARY OUTCOMES:
Adverse events | 30th minutes after
  30th minutes after the study drug administered

OTHER OUTCOMES:
Reduction in verbal rating scale | 15 minutes interval
  The pain of the study subjects was measured after 15th and 30th minutes later after the study drug administered.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Turkcuer, assoc. prof., Study Director — Pamukkale University
Locations (1):
- Pamukkale University Hospital, Emergency Department, Denizli, Turkey (Türkiye)

REFERENCES:
- [Background] Hewitt DJ, Martin V, Lipton RB, Brandes J, Ceesay P, Gottwald R, Schaefer E, Lines C, Ho TW. Randomized controlled study of telcagepant plus ibuprofen or acetaminophen in migraine. Headache. 2011 Apr;51(4):533-43. doi: 10.1111/j.1526-4610.2011.01860.x. PMID 21457238
- [Background] Prior MJ, Codispoti JR, Fu M. A randomized, placebo-controlled trial of acetaminophen for treatment of migraine headache. Headache. 2010 May;50(5):819-33. doi: 10.1111/j.1526-4610.2010.01638.x. Epub 2010 Mar 5. PMID 20236342
- [Derived] Turkcuer I, Serinken M, Eken C, Yilmaz A, Akdag O, Uyan E, Kiray C, Elicabuk H. Intravenous paracetamol versus dexketoprofen in acute migraine attack in the emergency department: a randomised clinical trial. Emerg Med J. 2014 Mar;31(3):182-5. doi: 10.1136/emermed-2013-203044. Epub 2014 Jan 6. PMID 24394884